CLINICAL TRIAL: NCT00336180
Title: Adolescent Drug and HIV Prevention in South Africa
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Edward A. Smith, Interim Director, Penn State University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01DA017491 (NIH); R01DA017491 (NIH)
Record Dates: First submitted 2006-06-09; First posted 2006-06-13 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Substance-Related Disorders; Sexually Transmitted Diseases
Keywords: Adolescent; Adolescent behavior; Adolescent development; Drinking behavior; Health behavior; Reproductive Behavior; Sexual Behavior; South Africa
MeSH Terms: conditions — Substance-Related Disorders; Sexually Transmitted Diseases; Adolescent Behavior; Drinking Behavior; Health Behavior; Reproductive Behavior; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HW (Experimental): The experimental group (HW) receives 18 classroom-based lessons on leisure motivation, life skills, and skills to avoid substance use and sexual risk.
  Interventions: Behavioral: HealthWise South Africa curriculum

INTERVENTIONS:
Behavioral: HealthWise South Africa curriculum — 18 classroom lessons

SUMMARY:
The purpose of this trial is to test the effectiveness of a classroom-based prevention program (HealthWise: Learning Life Skills for Young Adults) to reduce the risk of HIV/AIDS and STIs, as well as substance use, among adolescents in one area of South Africa.

DETAILED DESCRIPTION:
Recent estimates of the incidence of HIV among South African youth reveal rates to be among the highest in the world. Research shows that the sexual behaviors that put youth at increased risk for HIV often occur in the context of substance use. Consequently, effective prevention programs will most likely target both types of risk behavior. Research and theory also suggest that a positive youth development approach may be an useful way to reduce risk behavior. Therefore, our study involves the implementation of a classroom-based leisure, life-skill, and sexuality education curriculum, HealthWise: Learning Life Skills for Young Adults. This program is designed to reduce substance use and sexual risk behavior and to increase healthy leisure behavior and intra- and interpersonal skills.

Students from 4 high schools are currently receiving the HealthWise lessons in the 8th and 9th grades; students from 5 other schools serve as controls. Participants complete survey assessments on PalmPilots twice per year, until they leave school. Three cohorts of students are participating in this trial.

Our hypothesis is that HealthWise participants will engage in less risk behavior than controls. This will be tested using various statistical methodologies, including multiple regression, structural equation modeling, and growth modeling.

ELIGIBILITY:
Inclusion Criteria:

* attending one of nine secondary schools involved in the HealthWise South Africa research trial

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 7695 (Actual)
Dates: Start 2003-09; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
incidence of ATOD use | 2 years
incidence of lifetime sexual intercourse | 2 years
rates of condom use | 2 years
number of sexual partners | 2 years

SECONDARY OUTCOMES:
knowledge and attitudes about substances and sex | 2 years
healthy leisure attitudes/behaviors | 2 years
levels of inter- and intrapersonal skills | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Smith, DrPH, Principal Investigator — The Pennsylvania State University; Linda L Caldwell, PhD, Principal Investigator — The Pennsylvania State University
Locations (1):
- University of the Western Cape, Bellville, South Africa

REFERENCES:
- [Background] Caldwell L, Smith E, Wegner L, Vergnani T, Mpofu E, Flisher AJ, Mathews, C. HealthWise South Africa: Development of a life skills curriculum for young adults. World Leisure 3: 4-17, 2004.